CLINICAL TRIAL: NCT00540267
Title: Bone Mineral Density in the Korean Patients With Chronic Schizophrenia With Alcohol Abuse
Brief Title: Bone Density in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Joo Shim, Imje University Busan Paik Hospital
Other Study IDs: BMD07; Korea Health 21 R&D Project
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-10

CONDITIONS: Schizophrenia; Alcohol Abuse
Keywords: Schizophrenia; Alcohol Abuse; Bone Density
MeSH Terms: conditions — Schizophrenia; Alcoholism

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schizophrenia: Chronic schizophrenia with aged 18-80 years
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
People with chronic mental disorder such as schizophrenia and alcohol abuse are high risk groups for developing osteoporosis.

To evaluate the prevalence of bone mineral density in men patients with schizophrenia with alcohol abuse, the investigators will compare bone mineral density between patient with schizophrenia with and without alcohol abuse.

DETAILED DESCRIPTION:
People with schizophrenia has been known as a high risk groups for developing osteoporosis, because of lack of exercise, poor nutrition and high rate of smoking. Those with alcohol abuse may be higher risk group than one with schizophrenia without alcohol abuse, because they frequently have several medical problems such as liver dysfunction, Vitamin D deficiency, hyperparathyroidism and those medical condition increase risk for developing osteoporosis. Also alcohol itself can increase bone loss too by disturbing bone remodeling and enhancing bone fragility. To compare the prevalence of bone mineral density in patients with schizophrenia with alcohol abuse to those without alcohol problem, we will investigate BMD in large population of Korean patients with those illnesses.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia
* Onset of illness more than 5 years.

Exclusion Criteria:

* No severe Medical and endocrinological disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people with schizophrenia, gaed between 18-80 years, with no endocrine disorder
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The change of bone mineral density | cross sectional and prospective

SECONDARY OUTCOMES:
The effects of Smoking and antipsychotic drug on BMD | Cross sectional Study

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Cheol Shim, MD,PhD, Study Director — Inje University
Locations (1):
- Joo-Cheol Shim, Busan, South Korea